CLINICAL TRIAL: NCT02389946
Title: BIOTRONIK - A Prospective Randomized Multicenter Study to Assess the SaFety and Effectiveness of the Orsiro SiroLimus Eluting Coronary Stent System in the Treatment Of Subjects With up to Three De Novo or Restenotic Coronary Artery Lesions - V
Brief Title: Safety and Effectiveness of the Orsiro Sirolimus Eluting Coronary Stent System in Subjects With Coronary Artery Lesions
Acronym: BIOFLOW-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Collaborators: Biotronik AG (Industry); Baim Institute for Clinical Research (Other); Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOFLOW-V
Record Dates: First submitted 2015-03-02; First posted 2015-03-17 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease; Atherosclerosis, Coronary; Myocardial Ischemia; Ischemic Heart Disease; Acute Coronary Syndrome; Angina Pectoris
Keywords: Drug eluting coronary stents; Sirolimus; Bioabsorbable polymer; DES
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Angina Pectoris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orsiro sirolimus coronary stent system (Experimental): Intervention with a Orsiro DES.
  Interventions: Device: Orsiro DES
- Xience everolimus coronary stent system (Active Comparator): Intervention with a Xience DES.
  Interventions: Device: Xience DES

INTERVENTIONS:
Device: Orsiro DES — Orsiro is a device/drug combination product composed of two components, a device (coronary stent system including a cobalt chromium stent platform), and a drug product (a formulation of sirolimus) contained in a bioabsorbable polymer coating.
  Other Names: Orsiro sirolimus coronary stent system
  Arms: Orsiro sirolimus coronary stent system
Device: Xience DES
  Other Names: Xience everolimus coronary stent system
  Arms: Xience everolimus coronary stent system

SUMMARY:
The objective of this study is to assess the safety and efficacy of the Orsiro Sirolimus Eluting Coronary Stent System in the treatment of subjects with up to three native de novo or restenotic (standard PTCA only) coronary artery lesions compared to the Xience coronary stent system.

DETAILED DESCRIPTION:
The BIOTRONIK BIOFLOW-V clinical trial is a prospective, multicenter, randomized, controlled trial combining data on the randomized subjects with data from two historical studies by employing a Bayesian approach.

Subjects with CAD that qualify for PCI with stenting will be screened per the protocol inclusion and exclusion criteria to achieve a total of up to 1,400 randomized subjects. Eligible subjects will be randomized in a 2:1 ratio, stratified by study center, to undergo percutaneous coronary revascularization with either the Orsiro Sirolimus Eluting Stent System (treatment group) or the Xience Everolimus Eluting Stent System (control group).

Subjects may receive treatment of up to three target lesions, one or two target lesions per target vessel, for a maximum of two target vessels. The target lesion(s) must be de novo or restenotic lesion(s) of ≤ 36 mm in length in native coronary artery(ies), with a reference vessel diameter of 2.25-4.0 mm. Treatment of restenotic lesions is allowed provided that the target lesion was previously treated with PTCA only. All treatment with study stents is to be performed during a single index procedure. Note: Concurrent treatment of non-target lesions during the index procedure is not allowed.

Randomized subjects will have clinical follow-up at 1 month, 6 months, 12 months and at 2, 3, 4 and 5 years following the index procedure.

To assess the non-inferiority of the Orsiro stent compared to the Xience stent, BIOFLOW-V randomized subjects will be combined with historical subjects from the BIOFLOW-II and BIOFLOW-IV randomized trials employing a Bayesian approach. Only subjects who meet all clinical and angiographic eligibility criteria of the BIOFLOW-V trial will be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years or the minimum age required for legal adult consent in the country of enrollment.
2. Subject is an acceptable candidate for PCI.
3. Subject is an acceptable candidate for CABG.
4. Subject has clinical evidence of ischemic heart disease, stable or unstable angina pectoris or documented silent ischemia.
5. Subject is eligible for dual anti-platelet therapy treatment with aspirin plus either, clopidogrel, prasugrel, ticagrelor or ticlopidine.
6. Subject has provided written informed consent.
7. Subject is willing to comply with study follow-up requirements.

Each target lesion/vessel must meet all of the following angiographic criteria for the subject to be eligible for the trial:

1. Subject has up to three target lesions in up to two separate target vessels (two target lesions in one vessel and one target lesion in a separate vessel).
2. Target lesion must be de novo or restenotic lesion in native coronary artery; restenotic lesion must have been treated with a standard PTCA only.
3. Target lesion must be in major coronary artery or branch (target vessel).
4. Target lesion must have angiographic evidence of ≥ 50% and < 100% stenosis (by operator visual estimate). If the target lesion is < 70% stenosed, clinical evidence of ischemia by positive functional study, CT, electrocardiography, FFR, or post infarct angina.
5. TIMI flow > 1.
6. Target lesion must be ≤ 36 mm in length by operator visual estimate.
7. Target vessel RVD of 2.25-4.0 mm by operator visual estimate.
8. Target lesion must be treatable with a maximum of two overlapping stents.

Exclusion Criteria:

1. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation myocardial infarction (STEMI) within 72 hours prior to the index procedure. Hemodynamically stable non-STEMI (NSTEMI) subjects are eligible for study enrollment.
2. Subject is hemodynamically unstable.
3. Subject is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study.
4. Subject has a known allergy to contrast medium that cannot be adequately pre-medicated, or any known allergy to thienopyridine, aspirin, both heparin and bivalirudin, L-605 cobalt-chromium (Co-Cr) alloy or one of its major elements (cobalt, chromium, tungsten and nickel), acrylic, fluoropolymers, silicon carbide, PLLA, sirolimus or everolimus.
5. Revascularization of any target vessel within 9 months prior to the index procedure or previous PCI of any non-target vessel within 30 days prior to the index procedure.
6. Planned treatment of a lesion not meeting angiographic inclusion and exclusion criteria during the index procedure or after the index procedure.
7. Planned surgery within 6 months of index procedure unless dual antiplatelet therapy can be maintained throughout the peri-surgical period.
8. History of a stroke or transient ischemic attack (TIA) within 6 months prior to the index procedure.
9. Subjects with active bleeding disorders, active coagulopathy, or any other reason, who are ineligible for DAPT.
10. Subject will refuse blood transfusions.
11. Subject has documented left ventricular ejection fraction (LVEF) < 30% within 90 days prior to the index procedure.
12. Subject is dialysis-dependent.
13. Subject has impaired renal function (i.e., blood creatinine > 2.5 mg/dL or 221 μmol/L determined within 7 days prior to the index procedure).
14. Subject has leukopenia (i.e. < 3,000 white blood cells/mm3), thrombocytopenia (i.e. < 100,000 platelets/mm3) or thrombocytosis (i.e. > 700,000 platelet/mm3).
15. Subject is receiving oral or intravenous immunosuppressive therapy (inhaled steroids are permitted), or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus; diabetes mellitus is permitted).
16. Subject is receiving chronic anticoagulation (e.g. coumadin, dabigatran, apixaban, rivaroxaban or any other agent).
17. Subject has life expectancy of < 1 year.
18. Subject is participating in another investigational (medical device or drug) clinical study. Subjects may be concurrently enrolled in a post-market study, as long as the post-market study device, drug or protocol does not interfere with the investigational treatment or protocol of this study.
19. In the investigator's opinion, subject will not be able to comply with the follow-up requirements.

Subjects will be excluded from the trial if any of the target lesions/vessels meets any of the following angiographic criteria:

1. Target lesion is located within a saphenous vein graft or arterial graft.
2. Target lesion is a restenotic lesion that was previously treated with a bare metal or drug eluting stent (in-stent restenosis).
3. Target lesion has any of the following characteristics:

   1. Lesion location is within the left main coronary artery, or within 3 mm of the origin of the left anterior descending (LAD) or left circumflex (LCX).
   2. Involves a side branch of > 2.0 mm in diameter. Note: Lesions within 3 mm of the origin of the right coronary artery may be treated.
4. Target vessel/lesion is excessively tortuous/angulated or is severely calcified, that would prevent complete inflation of an angioplasty balloon. This assessment should be based on visual estimation.
5. Target vessel has angiographic evidence of thrombus.
6. Target lesion is totally occluded (100% stenosis).
7. Target vessel was treated with brachytherapy any time prior to the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1334 (Actual)
Dates: Start 2015-05; Primary Completion 2017-04 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Study Chair — Medstar Health Research Institute; David Kandzari, MD, Principal Investigator — Piedmont Heart Institute; Jacques Koolen, MD, Principal Investigator — Catharina Ziekenhuis
Locations (84):
- United States (52):
  - Fairhope, Alabama
  - Concord, California
  - La Mesa, California
  - Laguna Hills, California
  - Mission Viejo, California
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Hollywood, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Urbana, Illinois
  - Fort Wayne, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Bay City, Michigan
  - Detroit, Michigan
  - Lansing, Michigan
  - Pontiac, Michigan
  - Rochester, Michigan
  - Troy, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - Neptune City, New Jersey
  - Newark, New Jersey
  - New York, New York
  - Asheville, North Carolina
  - Greensboro, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Elyria, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Butler, Pennsylvania
  - Mechanicsburg, Pennsylvania
  - Wynnewood, Pennsylvania
  - York, Pennsylvania
  - Providence, Rhode Island
  - Greenville, South Carolina
  - Rock Hill, South Carolina
  - Knoxville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - McKinney, Texas
  - Tyler, Texas
  - Charlottesville, Virginia
  - Virginia Beach, Virginia
  - Charleston, West Virginia
- Adelaide, Australia
- Belgium (3):
  - Genk
  - Leuven
  - Roeselare
- Calgary, Alberta, Canada
- Aarhus, Denmark
- Germany (5):
  - Bad Segeberg
  - Berlin
  - Hamburg
  - Minden
  - Neuss
- Hungary (3):
  - Budapest
  - Pécs
  - Szeged
- Israel (5):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Rehovot
  - Tel Aviv
- Netherlands (3):
  - Breda
  - Eindhoven
  - Nieuwegein
- Auckland, New Zealand
- South Korea (3):
  - Daegu
  - Gwangju
  - Seoul
- Spain (4):
  - Barcelona
  - Madrid
  - Málaga
  - Seville
- Switzerland (2):
  - Lausanne
  - Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doros G, Massaro JM, Kandzari DE, Waksman R, Koolen JJ, Cutlip DE, Mauri L. Rationale of a novel study design for the BIOFLOW V study, a prospective, randomized multicenter study to assess the safety and efficacy of the Orsiro sirolimus-eluting coronary stent system using a Bayesian approach. Am Heart J. 2017 Nov;193:35-45. doi: 10.1016/j.ahj.2017.08.001. Epub 2017 Aug 5. PMID 29129253
- [Result] Kandzari DE, Mauri L, Koolen JJ, Massaro JM, Doros G, Garcia-Garcia HM, Bennett J, Roguin A, Gharib EG, Cutlip DE, Waksman R; BIOFLOW V Investigators. Ultrathin, bioresorbable polymer sirolimus-eluting stents versus thin, durable polymer everolimus-eluting stents in patients undergoing coronary revascularisation (BIOFLOW V): a randomised trial. Lancet. 2017 Oct 21;390(10105):1843-1852. doi: 10.1016/S0140-6736(17)32249-3. Epub 2017 Aug 26. PMID 28851504
- [Result] Kandzari DE, Koolen JJ, Doros G, Massaro JJ, Garcia-Garcia HM, Bennett J, Roguin A, Gharib EG, Cutlip DE, Waksman R; BIOFLOW V Investigators. Ultrathin Bioresorbable Polymer Sirolimus-Eluting Stents Versus Thin Durable Polymer Everolimus-Eluting Stents. J Am Coll Cardiol. 2018 Dec 25;72(25):3287-3297. doi: 10.1016/j.jacc.2018.09.019. Epub 2018 Sep 23. PMID 30257191
- [Result] Roguin A, Kandzari DE, Marcusohn E, Koolen JJ, Doros G, Massaro JM, Garcia-Garcia HM, Bennett J, Gharib EG, Cutlip DE, Waksman R. Subgroup Analysis Comparing Ultrathin, Bioresorbable Polymer Sirolimus-Eluting Stents Versus Thin, Durable Polymer Everolimus-Eluting Stents in Acute Coronary Syndrome Patients. Circ Cardiovasc Interv. 2018 Oct;11(10):e007331. doi: 10.1161/CIRCINTERVENTIONS.118.007331. PMID 30354631
- [Derived] Mankerious N, Toelg R, Abdelghani M, Garcia-Garcia HM, Farhan S, Allali A, Windecker S, Lefevre T, Saito S, Kandzari DE, Waksman R, Richardt G, Hemetsberger R. Impact of coronary artery tortuosity on outcomes following stenting with newer-generation drug-eluting stents. An analysis of the randomized BIOFLOW trials. Rev Esp Cardiol (Engl Ed). 2025 Aug;78(8):682-691. doi: 10.1016/j.rec.2024.12.009. Epub 2025 Jan 4. English, Spanish. PMID 39761745
- [Derived] Hemetsberger R, Mankerious N, Toelg R, Abdelghani M, Farhan S, Garcia-Garica HM, Allali A, Windecker S, Lefevre T, Saito S, Kandzari D, Waksman R, Richardt G. Patients with higher-atherothrombotic risk vs. lower-atherothrombotic risk undergoing coronary intervention with newer-generation drug-eluting stents: an analysis from the randomized BIOFLOW trials. Clin Res Cardiol. 2023 Sep;112(9):1278-1287. doi: 10.1007/s00392-023-02205-4. Epub 2023 Apr 16. PMID 37062047
- [Derived] Hemetsberger R, Abdelghani M, Toelg R, Garcia-Garcia HM, Farhan S, Mankerious N, Elbasha K, Allali A, Windecker S, Lefevre T, Saito S, Kandzari D, Waksman R, Richardt G. Complex vs. non-complex percutaneous coronary intervention with newer-generation drug-eluting stents: an analysis from the randomized BIOFLOW trials. Clin Res Cardiol. 2022 Jul;111(7):795-805. doi: 10.1007/s00392-022-01994-4. Epub 2022 Feb 25. PMID 35212802
- [Derived] Hemetsberger R, Abdelghani M, Toelg R, Mankerious N, Allali A, Garcia-Garcia HM, Windecker S, Lefevre T, Saito S, Slagboom T, Kandzari D, Koolen J, Waksman R, Richardt G. Impact of Coronary Calcification on Clinical Outcomes After Implantation of Newer-Generation Drug-Eluting Stents. J Am Heart Assoc. 2021 Jun 15;10(12):e019815. doi: 10.1161/JAHA.120.019815. Epub 2021 May 29. PMID 34056911
- [Derived] Dan K, Garcia-Garcia HM, Kolm P, Windecker S, Saito S, Kandzari DE, Waksman R. Comparison of Ultrathin, Bioresorbable-Polymer Sirolimus-Eluting Stents and Thin, Durable-Polymer Everolimus-Eluting Stents in Calcified or Small Vessel Lesions. Circ Cardiovasc Interv. 2020 Sep;13(9):e009189. doi: 10.1161/CIRCINTERVENTIONS.120.009189. Epub 2020 Sep 8. PMID 32895004
- [Derived] Toelg R, Slagboom T, Waltenberger J, Lefevre T, Saito S, Kandzari DE, Koolen J, Richardt G. Individual patient data analysis of the BIOFLOW study program comparing safety and efficacy of a bioresorbable polymer sirolimus eluting stent to a durable polymer everolimus eluting stent. Catheter Cardiovasc Interv. 2021 Nov 1;98(5):848-856. doi: 10.1002/ccd.29254. Epub 2020 Sep 5. PMID 32890442
- [Derived] Kandzari DE, Koolen JJ, Doros G, Garcia-Garcia HM, Bennett J, Roguin A, Gharib EG, Cutlip DE, Waksman R; BIOFLOW V Investigators. Ultrathin Bioresorbable-Polymer Sirolimus-Eluting Stents Versus Thin Durable-Polymer Everolimus-Eluting Stents for Coronary Revascularization: 3-Year Outcomes From the Randomized BIOFLOW V Trial. JACC Cardiovasc Interv. 2020 Jun 8;13(11):1343-1353. doi: 10.1016/j.jcin.2020.02.019. PMID 32499026
- [Derived] Mattke S, Hanson M, Bentele M, Kandzari DE. Cost and Mortality Implications of Lower Event Rates After Implantation of an Ultrathin-Strut Coronary Stent Compared With a Thin-Strut Stent Over Four Years. Cardiovasc Revasc Med. 2020 Jul;21(7):835-842. doi: 10.1016/j.carrev.2019.12.018. Epub 2019 Dec 18. PMID 31954661
- [Derived] Mattke S, Hanson M, Dallmann AC, Bentele M. Health Economic Evaluation of an Ultrathin, Bioresorbable-Polymer Sirolimus-Eluting Coronary Stent Compared to a Thin, Durable-Polymer Everolimus-Eluting Stent. Cardiovasc Revasc Med. 2019 Sep;20(9):752-757. doi: 10.1016/j.carrev.2018.11.006. Epub 2018 Nov 20. PMID 30638888

RESULTS

PARTICIPANT FLOW:
Groups:
- Xience Everolimus Coronary Stent System: Intervention with a Xience DES.
  Xience DES
Period: Overall Study
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Started | 884 | 450
Completed | 860 | 435
Not Completed | 24 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System | Total
Number analyzed (Participants) | 884 | 450 | 1334
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (10.32) | 64.6 (10.67) | 64.5 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 122 | 346
  Male | 660 | 328 | 988
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 13 | 48
  Not Hispanic or Latino | 812 | 417 | 1229
  Unknown or Not Reported | 37 | 20 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 29 | 13 | 42
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 24 | 13 | 37
  White | 792 | 406 | 1198
  More than one race | 11 | 1 | 12
  Unknown or Not Reported | 27 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Target Lesion Failure (TLF) at 12 Months Post-Index Procedure by Bayesian Estimation
Description: TLF is defined as all cardiac death, target vessel Q-wave or non-Q-wave myocardial infarction (MI), or clinically driven target lesion revascularization (TLR).
Time Frame: 12-Months
Population: Pre-specified Bayesian analysis: BIOFLOW-V intent-to-treat subjects who experienced the primary endpoint or had at least 330 days of follow-up and BIOFLOW-II (NCT01356888) and BIOFLOW-IV (NCT01939249) subjects who satisfied the BIOFLOW-V inclusion/exclusion criteria and experienced the primary endpoint or had at least 330 days of follow-up.
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 883 | 427
Percentage of participants | 6.32 (0.75) | 8.90 (1.22)
Statistical Analysis 1: Comparison: Orsiro Sirolimus Coronary Stent System vs Xience Everolimus Coronary Stent System; Bayesian calculation using a hierarchical model to incorporate data from previous BIOFLOW-II and BIOFLOW-IV trials; Test type: Non-Inferiority — Non-inferiority of the 12-month TLF rate for the Orsiro stent vs. the Xience stent was assessed as the primary endpoint. The null hypothesis H0 was that the Orsiro stent would have a primary endpoint (12-month TLF) rate equal to or exceeding that of the Xience group by the non-inferiority margin or more. The alternative hypothesis HA was that the Orsiro stent would have a 12-month TLF rate less than the Xience group rate plus the non-inferiority margin of 3.85%; Posterior Probability of non-inferioriry = 100

2. Secondary Outcome: Number of Lesions With Device Success
Description: Defined as attainment of < 30% residual stenosis of the target lesion using the assigned study stent only.
Time Frame: Hospital Discharge (6-24 hours post-index procedure)
Population: Device Success per lesion. Lesions that were not treated and lesions missing both site-reported and core lab-assessed percent residual stenosis were excluded from the analysis.
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 881 | 445
Number analyzed (Lesions) | 1107 | 583
Lesions | 1082 | 566
Statistical Analysis 1: Comparison: Orsiro Sirolimus Coronary Stent System vs Xience Everolimus Coronary Stent System; Test type: Other; p = 0.415, Fisher Exact

3. Secondary Outcome: Number of Lesions With Lesion Success
Description: Defined as attainment of < 30% residual stenosis of the target lesion using any percutaneous method.
Time Frame: Hospital Discharge (6-24 hours post-index procedure)
Population: Lesion Success per lesion. Lesions that were not treated and lesions missing both site-reported and core lab-assessed percent residual stenosis were excluded from the analysis.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 881 | 445
Number analyzed (Lesions) | 1107 | 583
Lesions | 1102 | 579

4. Secondary Outcome: Number of Participants With Procedure Success
Description: Defined as attainment of < 30% residual stenosis of the target lesion using the assigned study stent only without occurrence of in-hospital major adverse cardiac events (MACE; composite of all-cause death, Q-wave or non-Q-wave MI, and any clinically-driven TLR).
Time Frame: Hospital Discharge (6-24 hours post-index procedure)
Population: Procedure success was analyzed per subject: for a subject to be considered a procedure success, all of the subject's target lesions had to be considered device success. Lesions that were not treated and lesions missing both site-reported and core lab-assessed percent residual stenosis were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 881 | 445
Participants | 827 | 401

5. Secondary Outcome: Number of Participants With Myocardial Infarction
Time Frame: Hospital Discharge (6-24 hours post-index procedure), 1, 6, 12 months, 2, 3, 4 and 5 years
Population: Analysis population for each outcome measure time frame is based on participants completing or experiencing an event at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 882 | 449
Participants
  6-24 hours post-index procedure | 34 | 30
  1-month post-index procedure: number analyzed (Participants) | 878 | 448
  1-month post-index procedure | 38 | 31
  6-month: number analyzed (Participants) | 865 | 442
  6-month | 40 | 36
  12-month: number analyzed (Participants) | 832 | 425
  12-month | 41 | 37
  2-year: number analyzed (Participants) | 831 | 419
  2-year | 56 | 42
  3-year: number analyzed (Participants) | 816 | 411
  3-year | 60 | 49
  4-year: number analyzed (Participants) | 792 | 404
  4-year | 66 | 52
  5-year: number analyzed (Participants) | 768 | 395
  5-year | 76 | 58

6. Secondary Outcome: Number of Participants With Myocardial Infarction or Cardiac Death
Time Frame: Hospital Discharge (6-24 hours post-index procedure), 1, 6, 12 months, 2, 3, 4 and 5 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 883 | 449
Participants
  Hospital Discharge (6-24 hours post-index procedure) | 35 | 30
  1-month: number analyzed (Participants) | 879 | 448
  1-month | 39 | 31
  6-month: number analyzed (Participants) | 866 | 442
  6-month | 41 | 37
  12-month: number analyzed (Participants) | 833 | 427
  12-month | 42 | 39
  2-year: number analyzed (Participants) | 836 | 420
  2-year | 61 | 43
  3-year: number analyzed (Participants) | 823 | 413
  3-year | 68 | 51
  4-year: number analyzed (Participants) | 808 | 406
  4-year | 82 | 54
  5-year: number analyzed (Participants) | 786 | 398
  5-year | 94 | 61

7. Secondary Outcome: Number of Participants With MACE and Individual MACE Components
Description: MACE events are defined as all-cause death, Q-wave or non-Q-wave MI, or any clinically-driven TLR. The number of participants with any MACE event is provided, as well as number of participants with each of the individual components.
Time Frame: Hospital Discharge (6-24 hours post-index procedure), 1, 6, 12 months, 2, 3, 4 and 5 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 883 | 449
Participants
  6-24 hours post-index MACE Total | 35 | 31
  6-24 hours post-index MACE Component: Death | 1 | 1
  6-24 hours post-index MACE Component: Protocol defined Q-Wave or non-Q-wave MI: number analyzed (Participants) | 882 | 449
  6-24 hours post-index MACE Component: Protocol defined Q-Wave or non-Q-wave MI | 34 | 30
  6-24 hours post-index MACE Component: Clinically-driven TLR: number analyzed (Participants) | 882 | 449
  6-24 hours post-index MACE Component: Clinically-driven TLR | 2 | 2
  1-month MACE Total: number analyzed (Participants) | 879 | 448
  1-month MACE Total | 39 | 32
  1-month MACE Component: Death: number analyzed (Participants) | 879 | 448
  1-month MACE Component: Death | 1 | 1
  1-month MACE Component: Protocol defined Q-Wave or non-Q-wave MI: number analyzed (Participants) | 878 | 448
  1-month MACE Component: Protocol defined Q-Wave or non-Q-wave MI | 38 | 31
  1-month MACE Component: Clinically-driven TLR: number analyzed (Participants) | 878 | 448
  1-month MACE Component: Clinically-driven TLR | 4 | 3
  6-month MACE Total: number analyzed (Participants) | 871 | 444
  6-month MACE Total | 53 | 42
  6-month MACE Component: Death: number analyzed (Participants) | 870 | 443
  6-month MACE Component: Death | 6 | 4
  6-month MACE Component: Protocol-defined Q-Wave or non-Q-wave MI: number analyzed (Participants) | 865 | 442
  6-month MACE Component: Protocol-defined Q-Wave or non-Q-wave MI | 40 | 36
  6-month MACE Component: Clinically-driven TLR: number analyzed (Participants) | 865 | 440
  6-month MACE Component: Clinically-driven TLR | 13 | 8
  12-month MACE Total: number analyzed (Participants) | 839 | 429
  12-month MACE Total | 59 | 44
  12-month MACE Component: Death: number analyzed (Participants) | 837 | 428
  12-month MACE Component: Death | 7 | 6
  12-month MACE Component: Protocol-defined Q-Wave or non-Q-wave MI: number analyzed (Participants) | 832 | 425
  12-month MACE Component: Protocol-defined Q-Wave or non-Q-wave MI | 41 | 37
  12-month MACE Component: Clinically-driven TLR: number analyzed (Participants) | 832 | 422
  12-month MACE Component: Clinically-driven TLR | 17 | 10
  2-year MACE Total: number analyzed (Participants) | 848 | 427
  2-year MACE Total | 85 | 56
  2-year MACE Component: Death: number analyzed (Participants) | 841 | 424
  2-year MACE Component: Death | 16 | 9
  2-year MACE Component: Protocol-defined Q-Wave or non-Q-wave MI: number analyzed (Participants) | 831 | 419
  2-year MACE Component: Protocol-defined Q-Wave or non-Q-wave MI | 56 | 42
  2-year MACE Component: Clinically-driven TLR: number analyzed (Participants) | 829 | 417
  2-year MACE Component: Clinically-driven TLR | 21 | 19
  3-year MACE Total: number analyzed (Participants) | 841 | 425
  3-year MACE Total | 102 | 73
  3-year MACE Component: Death: number analyzed (Participants) | 834 | 422
  3-year MACE Component: Death | 27 | 17
  3-year MACE Component: Protocol-defined Q-Wave or non-Q-wave MI: number analyzed (Participants) | 816 | 411
  3-year MACE Component: Protocol-defined Q-Wave or non-Q-wave MI | 60 | 49
  3-year MACE Component: Clinically-driven TLR: number analyzed (Participants) | 814 | 407
  3-year MACE Component: Clinically-driven TLR | 27 | 25
  4-year MACE Total: number analyzed (Participants) | 834 | 422
  4-year MACE Total | 133 | 81
  4-year MACE Component: Death: number analyzed (Participants) | 827 | 419
  4-year MACE Component: Death | 45 | 22
  4-year MACE Component: Protocol-defined Q-Wave or non-Q-wave MI: number analyzed (Participants) | 792 | 404
  4-year MACE Component: Protocol-defined Q-Wave or non-Q-wave MI | 66 | 52
  4-year MACE Component: Clinically-driven TLR: number analyzed (Participants) | 790 | 400
  4-year MACE Component: Clinically-driven TLR | 38 | 28
  5-year MACE Total: number analyzed (Participants) | 820 | 416
  5-year MACE Total | 155 | 92
  5-year MACE Component: Death: number analyzed (Participants) | 808 | 411
  5-year MACE Component: Death | 56 | 27
  5-year MACE Component: Protocol-defined Q-Wave or non-Q-wave MI: number analyzed (Participants) | 768 | 395
  5-year MACE Component: Protocol-defined Q-Wave or non-Q-wave MI | 76 | 58
  5-year MACE Clinically-driven TLR: number analyzed (Participants) | 761 | 388
  5-year MACE Clinically-driven TLR | 48 | 32

8. Secondary Outcome: Number of Participants With TLF and Individual TLF Components
Description: TLF events are defined as cardiac death, target vessel Q-wave or non-Q-wave MI, or any clinically-driven TLR. The number of participants with any TLF event is provided, as well as number of participants with each of the individual components.
Time Frame: Hospital Discharge (6-24 hours post-index procedure), 1, 6, 12 months, 2, 3, 4 and 5 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 883 | 449
Participants
  6-24 hours post-index TLF Total | 35 | 31
  6-24 hours post-index TLF Component: Cardiac Death | 1 | 1
  6-24 hours post-index TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 882 | 449
  6-24 hours post-index TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 34 | 29
  6-24 hours post-index TLF Component: Clinically-driven TLR: number analyzed (Participants) | 882 | 449
  6-24 hours post-index TLF Component: Clinically-driven TLR | 2 | 2
  1-month TLF Total: number analyzed (Participants) | 879 | 448
  1-month TLF Total | 37 | 32
  1-month TLF Component: Cardiac Death: number analyzed (Participants) | 879 | 448
  1-month TLF Component: Cardiac Death | 1 | 1
  1-month TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 878 | 448
  1-month TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 36 | 30
  1-month TLF Component: Clinically-driven TLR: number analyzed (Participants) | 878 | 448
  1-month TLF Component: Clinically-driven TLR | 4 | 3
  6-month TLF Total: number analyzed (Participants) | 866 | 442
  6-month TLF Total | 47 | 39
  6-month TLF Component: Cardiac Death: number analyzed (Participants) | 865 | 441
  6-month TLF Component: Cardiac Death | 1 | 2
  6-month TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 865 | 441
  6-month TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 38 | 34
  6-month TLF Component: Clinically-driven TLR: number analyzed (Participants) | 865 | 440
  6-month TLF Component: Clinically-driven TLR | 13 | 8
  12-month TLF Total: number analyzed (Participants) | 833 | 427
  12-month TLF Total | 52 | 41
  12-month TLF Component: Cardiac Death: number analyzed (Participants) | 831 | 425
  12-month TLF Component: Cardiac Death | 1 | 3
  12-month TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 831 | 424
  12-month TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 39 | 35
  12-month TLF Component: Clinically-driven TLR: number analyzed (Participants) | 832 | 422
  12-month TLF Component: Clinically-driven TLR | 17 | 10
  2-year TLF Total: number analyzed (Participants) | 836 | 421
  2-year TLF Total | 64 | 48
  2-year TLF Component: Cardiac Death: number analyzed (Participants) | 830 | 417
  2-year TLF Component: Cardiac Death | 5 | 2
  2-year TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 829 | 418
  2-year TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 45 | 39
  2-year TLF Component: Clinically-driven TLR: number analyzed (Participants) | 829 | 417
  2-year TLF Component: Clinically-driven TLR | 21 | 19
  3-year TLF Total: number analyzed (Participants) | 824 | 414
  3-year TLF Total | 72 | 56
  3-year TLF Component: Cardiac Death: number analyzed (Participants) | 817 | 410
  3-year TLF Component: Cardiac Death | 9 | 5
  3-year TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 814 | 409
  3-year TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 46 | 41
  3-year TLF Component: Clinically-driven TLR: number analyzed (Participants) | 814 | 407
  3-year TLF Component: Clinically-driven TLR | 27 | 25
  4-year TLF Total: number analyzed (Participants) | 809 | 407
  4-year TLF Total | 91 | 60
  4-year TLF Component: Cardiac Death: number analyzed (Participants) | 801 | 403
  4-year TLF Component: Cardiac Death | 17 | 5
  4-year TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 790 | 402
  4-year TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 49 | 44
  4-year TLF Component: Clinically-driven TLR: number analyzed (Participants) | 790 | 400
  4-year TLF Component: Clinically-driven TLR | 38 | 28
  5-year TLF Total: number analyzed (Participants) | 787 | 399
  5-year TLF Total | 104 | 66
  5-year TLF Component: Cardiac Death: number analyzed (Participants) | 774 | 392
  5-year TLF Component: Cardiac Death | 21 | 8
  5-year TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 765 | 391
  5-year TLF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 56 | 45
  5-year TLF Component: Clinically-driven TLR: number analyzed (Participants) | 761 | 388
  5-year TLF Component: Clinically-driven TLR | 48 | 32

9. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) and Individual TVF Components
Description: TVF events are defined as cardiac death, target vessel Q-wave or non-Q-wave MI, or any clinically-driven TVR. The number of participants with any TVF event is provided, as well as number of participants with each of the individual components.
Time Frame: Hospital Discharge (6-24 hours post-index procedure), 1, 6, 12 months, 2, 3, 4 and 5 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 883 | 449
Participants
  6-24 hours post-index TVF Total | 35 | 31
  6-24 hours post-index TVF Component: Cardiac Death | 1 | 1
  6-24 hours post-index TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 882 | 449
  6-24 hours post-index TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 34 | 29
  6-24 hours post-index TVF Component: Clinically-driven TVR: number analyzed (Participants) | 882 | 449
  6-24 hours post-index TVF Component: Clinically-driven TVR | 2 | 2
  1-month TVF Total: number analyzed (Participants) | 879 | 448
  1-month TVF Total | 38 | 32
  1-month TVF Component: Cardiac Death: number analyzed (Participants) | 879 | 448
  1-month TVF Component: Cardiac Death | 1 | 1
  1-month TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 878 | 448
  1-month TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 36 | 30
  1-month TVF Component: Clinically-driven TVR: number analyzed (Participants) | 878 | 448
  1-month TVF Component: Clinically-driven TVR | 5 | 4
  6-month TVF Total: number analyzed (Participants) | 866 | 442
  6-month TVF Total | 51 | 40
  6-month TVF Component: Cardiac Death: number analyzed (Participants) | 865 | 441
  6-month TVF Component: Cardiac Death | 1 | 2
  6-month TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 865 | 441
  6-month TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 38 | 34
  6-month TVF Component: Clinically-driven TVR: number analyzed (Participants) | 865 | 440
  6-month TVF Component: Clinically-driven TVR | 18 | 10
  12-month TVF Total: number analyzed (Participants) | 834 | 427
  12-month TVF Total | 60 | 45
  12-month TVF Component: Cardiac Death: number analyzed (Participants) | 831 | 425
  12-month TVF Component: Cardiac Death | 1 | 3
  12-month TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 831 | 424
  12-month TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 39 | 35
  12-month TVF Component: Clinically-driven TVR: number analyzed (Participants) | 833 | 422
  12-month TVF Component: Clinically-driven TVR | 27 | 15
  2-year TVF Total: number analyzed (Participants) | 836 | 422
  2-year TVF Total | 74 | 56
  2-year TVF Component: Cardiac Death: number analyzed (Participants) | 830 | 417
  2-year TVF Component: Cardiac Death | 5 | 2
  2-year TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 829 | 418
  2-year TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 45 | 39
  2-year TVF Component: Clinically-driven TVR: number analyzed (Participants) | 829 | 418
  2-year TVF Component: Clinically-driven TVR | 37 | 30
  3-year TVF Total: number analyzed (Participants) | 824 | 415
  3-year TVF Total | 84 | 68
  3-year TVF Component: Cardiac Death: number analyzed (Participants) | 817 | 410
  3-year TVF Component: Cardiac Death | 9 | 5
  3-year TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 814 | 409
  3-year TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 46 | 41
  3-year TVF Component: Clinically-driven TVR: number analyzed (Participants) | 814 | 408
  3-year TVF Component: Clinically-driven TVR | 45 | 40
  4-year TVF Total: number analyzed (Participants) | 809 | 409
  4-year TVF Total | 110 | 74
  4-year TVF Component: Cardiac Death: number analyzed (Participants) | 801 | 403
  4-year TVF Component: Cardiac Death | 17 | 5
  4-year TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 790 | 402
  4-year TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 49 | 44
  4-year TVF Component: Clinically-driven TVR: number analyzed (Participants) | 790 | 402
  4-year TVF Component: Clinically-driven TVR | 63 | 46
  5-year TVF Total: number analyzed (Participants) | 788 | 401
  5-year TVF Total | 127 | 81
  5-year TVF Component: Cardiac Death: number analyzed (Participants) | 774 | 392
  5-year TVF Component: Cardiac Death | 21 | 8
  5-year TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI: number analyzed (Participants) | 765 | 391
  5-year TVF Component: Protocol-defined Target Vessel Q-wave or non-Q-Wave MI | 56 | 45
  5-year TVF Component: Clinically-driven TVR: number analyzed (Participants) | 763 | 390
  5-year TVF Component: Clinically-driven TVR | 78 | 51

10. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: Stent thrombosis according to the Academic Research Consortium criteria.
Time Frame: 24 hours, 30 days, 1 year, and 5 years post-index procedure
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
Number analyzed (Participants) | 884 | 450
Participants
  Possible ARC Stent Thrombosis Total: number analyzed (Participants) | 764 | 390
  Possible ARC Stent Thrombosis Total | 11 | 6
  Possible ARC Stent Thrombosis Acute (<=24 hours) | 0 | 0
  Possible ARC Stent Thrombosis Sub-acute (>24 hours and <=30 days): number analyzed (Participants) | 879 | 449
  Possible ARC Stent Thrombosis Sub-acute (>24 hours and <=30 days) | 0 | 0
  Possible ARC Stent Thrombosis Late (>30 days and <=1 year): number analyzed (Participants) | 753 | 385
  Possible ARC Stent Thrombosis Late (>30 days and <=1 year) | 0 | 1
  Possible ARC Stent Thrombosis Very Late (>1 year): number analyzed (Participants) | 764 | 389
  Possible ARC Stent Thrombosis Very Late (>1 year) | 11 | 5
  Definite/Probable ARC Stent Thrombosis Total: number analyzed (Participants) | 756 | 385
  Definite/Probable ARC Stent Thrombosis Total | 5 | 7
  Definite/Probable ARC Stent Thrombosis Acute (<=24 hours) | 1 | 0
  Definite/Probable ARC Stent Thrombosis Sub-acute (>24 hours and <=30 days): number analyzed (Participants) | 879 | 449
  Definite/Probable ARC Stent Thrombosis Sub-acute (>24 hours and <=30 days) | 2 | 1
  Definite/Probable ARC Stent Thrombosis Late (>30 days and <=1 year): number analyzed (Participants) | 753 | 384
  Definite/Probable ARC Stent Thrombosis Late (>30 days and <=1 year) | 1 | 2
  Definite/Probable ARC Stent Thrombosis Very Late (>1 year): number analyzed (Participants) | 753 | 384
  Definite/Probable ARC Stent Thrombosis Very Late (>1 year) | 1 | 4

ADVERSE EVENTS:
Time Frame: 5 year
Arm/Group | Orsiro Sirolimus Coronary Stent System | Xience Everolimus Coronary Stent System
All-Cause Mortality (participants affected / at risk) | 56/884 | 27/450
Serious Adverse Events (participants affected / at risk) | 548/884 | 293/450
Other Adverse Events (participants affected / at risk) | 291/884 | 165/450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orsiro Sirolimus Coronary Stent System (N=884) | Xience Everolimus Coronary Stent System (N=450)
Anaemia (Blood and lymphatic system disorders) | 11 (12) | 5 (5)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 6 (7) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 46 (58) | 24 (33)
Angina pectoris (Cardiac disorders) | 85 (105) | 49 (61)
Angina unstable (Cardiac disorders) | 53 (64) | 32 (43)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 2 (6)
Atrial fibrillation (Cardiac disorders) | 36 (48) | 18 (26)
Atrial flutter (Cardiac disorders) | 7 (8) | 4 (4)
Atrial tachycardia (Cardiac disorders) | 2 (5) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 1 (1)
Bradycardia (Cardiac disorders) | 7 (7) | 4 (5)
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 20 (36) | 10 (14)
Cardiac failure (Cardiac disorders) | 15 (17) | 5 (5)
Cardiac pseudoaneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 3 (3) | 1 (1)
Coronary artery disease (Cardiac disorders) | 16 (23) | 13 (16)
Coronary artery dissection (Cardiac disorders) | 23 (24) | 20 (22)
Coronary artery embolism (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 11 (13) | 10 (10)
Coronary artery stenosis (Cardiac disorders) | 115 (205) | 58 (121)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 6 (6) | 7 (7)
Myocardial rupture (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (2)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 3 (4)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 2 (3) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 6 (8) | 3 (4)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 11 (17) | 4 (4)
Retinal detachment (Eye disorders) | 3 (3) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 2 (2)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (15) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal angina (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 4 (6) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 4 (9) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (5) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 6 (8) | 0 (0)
Stomach granuloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Accidental death (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (6) | 3 (3)
Catheter site haematoma (General disorders) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 22 (25) | 6 (6)
Death (General disorders) | 8 (8) | 2 (2)
Incarcerated hernia (General disorders) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 92 (121) | 41 (61)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Vascular stent restenosis (General disorders) | 24 (27) | 14 (15)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (2) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Serum sickness (Immune system disorders) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 2 (3) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4) | 1 (1)
Catheter site abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 8 (13) | 4 (4)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Emphysematous cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (3) | 2 (2)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 29 (31) | 10 (15)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 13 (14) | 9 (10)
Septic shock (Infections and infestations) | 4 (4) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (3) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 15 (18) | 6 (6)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 2 (2) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Asbestosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Femur fracture (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 3 (3) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 3 (3) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (5) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 (20) | 11 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 3 (3)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 3 (4)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 2 (3) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 8 (8) | 4 (5)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (3) | 5 (7)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 9 (9) | 4 (4)
Embolic stroke (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 4 (5) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Presyncope (Nervous system disorders) | 6 (6) | 1 (1)
Syncope (Nervous system disorders) | 20 (21) | 7 (7)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 4 (5) | 4 (4)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 3 (3)
Confusional state (Psychiatric disorders) | 3 (3) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 4 (4)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 21 (30) | 11 (17)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 2 (3)
Chronic kidney disease (Renal and urinary disorders) | 12 (12) | 3 (3)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 6 (10) | 3 (3)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal mass (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 6 (6) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 (26) | 9 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (33) | 11 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 6 (7)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diffuse cutaneous mastocytosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 7 (7) | 2 (2)
Femoral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 6 (6)
Hypertensive crisis (Vascular disorders) | 7 (8) | 1 (2)
Hypotension (Vascular disorders) | 7 (7) | 5 (5)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 4 (6) | 4 (6)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 8 (9) | 4 (5)
Peripheral artery stenosis (Vascular disorders) | 10 (11) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 5 (5) | 3 (3)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 2 (2) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anginal equivalent (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 3 (3) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 2 (2) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 4 (4) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 3 (3) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Necrotising retinitis (Eye disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 1 (1)
Retinal artery embolism (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal polyp (Gastrointestinal disorders) | 3 (3) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Cyst (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 6 (6) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (3) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Picornavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 3 (3)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incomplete spinal fusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Carotid bruit (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevaction (Investigations) | 1 (1) | 0 (0)
Scan myocardial perfusion abnormal (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Deformity thorax (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neuroendocrine tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (11)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
Urethral cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amyotropic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 2 (2) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 4 (4)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 3 (3) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy idiopathic progressive (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 3 (3) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosomatic disease (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 0 (0) | 2 (2)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 1 (1)
Brachiocephalic artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (6) | 2 (2)
Femoral artery occlusion (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Labile hypertension (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
May-Thurner syndrome (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 6 (6) | 1 (1)
Penetrating aortic ulcer (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Steal syndrome (Vascular disorders) | 1 (1) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orsiro Sirolimus Coronary Stent System (N=884) | Xience Everolimus Coronary Stent System (N=450)
Angina pectoris (Cardiac disorders) | 159 (215) | 94 (125)
Non-cardiac chest pain (General disorders) | 163 (240) | 89 (128)
Myocardial necrosis marker increased (Investigations) | 174 (176) | 90 (91)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 100 (112) | 45 (52)
Acute Myocardial Infarction (Cardiac disorders) | 49 (61) | 26 (35)
Angina Unstable (Cardiac disorders) | 67 (89) | 40 (54)
Atrial Fibrillation (Cardiac disorders) | 60 (75) | 27 (38)
Coronary Artery Dissection (Cardiac disorders) | 32 (33) | 24 (26)
Coronary Artery Stenosis (Cardiac disorders) | 120 (215) | 61 (126)
Fatigue (General disorders) | 36 (36) | 25 (25)
Dizziness (Nervous system disorders) | 51 (51) | 21 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02389946/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT02389946/SAP_001.pdf